CLINICAL TRIAL: NCT01211184
Title: Fluid and Nutrition in Elective Hip Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sodertalje Hospital (Other)
Responsible Party: Principal Investigator, Robert Hahn, Research Director, Sodertalje Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STS1
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Results first posted 2011-12-13 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-10

CONDITIONS: Hip Surgery Corrective
Keywords: Hip surgery; Metabolism; Glucose; Body fluids; Complications
MeSH Terms: interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fasting (Placebo Comparator): patients undergo surgery in the fasting state
  Interventions: Behavioral: Fasting.
- Water administration (Active Comparator): Patients undergo hip surgery after receiving 800 ml water by mouth the morning 2 hours before surgery
  Interventions: Dietary Supplement: Water administration
- carbohydrate drink (Active Comparator): Patients undergo hip surgery after receiving 800 ml carbohydrate drink by mouth
  Interventions: Dietary Supplement: carbohydrate drink

INTERVENTIONS:
Dietary Supplement: Water administration — patients undergo hip surgery after receiving 800 ml water by mouth in the morning before the surgery.
  Other Names: Tap water
  Arms: Water administration
Dietary Supplement: carbohydrate drink — 800 ml carbohydrate drink by mouth the evening before surgery and 400 ml carbohydrate drink by mouth 2 hours before surgery
  Other Names: PreOp Nutricia ( Nutricia Nordic AB)
  Arms: carbohydrate drink
Behavioral: Fasting. — The patient is fasting from midnight before the surgery.
  Arms: Fasting

SUMMARY:
The purpose of this study is to determine whether fluid or glucose administration before hip replacement surgery minimizes postoperative muscle breakdown (catabolism), fatigue and disturbances in carbohydrate metabolism.

DETAILED DESCRIPTION:
1. How can a simple and safe way to measure the body's tendency to transient diabetes associated with surgery?
2. Can fluid or glucose administration before elective hip surgery, minimizing post-operative muscle breakdown (catabolism), fatigue and disturbances in carbohydrate metabolism?

ELIGIBILITY:
Inclusion Criteria: Patient scheduled for hip surgery. Exclusion Criteria: Endocrinological disorders.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Hahn, Prof, Study Chair — Linkoeping University
Locations (1):
- Södertälje Hospital, Södertälje, Södertälje, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Results have been published in international journals. Main article is:
  Ljunggren S, Hahn RG. Oral nutrition or water loading before hip replacement surgery; a randomized clinical trial. Trials 2012; 13: 97.

REFERENCES:
- [Derived] Ljunggren S, Hahn RG. Oral nutrition or water loading before hip replacement surgery; a randomized clinical trial. Trials. 2012 Jul 2;13:97. doi: 10.1186/1745-6215-13-97. PMID 22747890

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 patients were recruited from the Department of Orthopedics between May 2008 and September 2009
Pre-assignment Details: Information about the study, exclusion criteriae were applied to potential subjects
Groups:
- Water: Patients undergo hip surgery after receiving 800 ml water by mouth the evening before surgery
Period: Overall Study
Arm/Group | Fasting | Water | Carbohydrate Drink
Started | 20 | 20 | 20
Completed | 20 | 18 | 19
Not Completed | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fasting | Water | Carbohydrate Drink | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 11 | 25
  >=65 years | 13 | 13 | 9 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (9.6) | 66.4 (10.6) | 65.2 (8.0) | 66.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 12 | 42
  Male | 3 | 7 | 8 | 18
Region of Enrollment [Number; unit: participants]
  Sweden | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Sensitivity (Percent)
Description: Insulin sensitivity (micro-mol per kg per minute glucose uptake) was calculated based on an intravenous glucose tolerance test (Theor Biol Med Model 2011, 8: 12) on the day before surgery. The percent change was taken as (day after - day before) / day before
Time Frame: Day before surgery (approximately 3 PM) and in the morning after surgery (approx. 7.30 AM).
Population: Per protocol analysis. The study was powered to detect a difference in glucose clearance.
Measure: Median (Inter-Quartile Range); unit: percent change of insulin sensitivity
Groups:
- Fasting Group: Patients did not ingest any drink or food from midnight before the surgery.
- Water Group: Patients drank 800 ml of tap water 2 hrs before entering the operating room
- Nutrition Group: Patients drank 800 ml in the evening before surgery and 400 ml 2 hours before surgery of a commercially available carbohydrate drink (PreOp)
Arm/Group | Fasting Group | Water Group | Nutrition Group
Number analyzed (Participants) | 16 | 14 | 15
percent change of insulin sensitivity | -43 [-77 to 19] | -38 [-82 to -20] | -51 [-74 to 0]

2. Secondary Outcome: Muscle Catabolism
Description: Assessed by the ratio of 3-methylhistidine/creatinine in excreted urine (unit: mmol/mmol).This is an amino acid unique to muscle that does not undergo intermediary metabolism, meaning that its urinary excretion is an index of the degree of muscle catabolism.
Time Frame: From the morning after surgery (07.30) up to the morning two days after sthe surgery (07.30)
Population: Per protocol
Measure: Mean (Standard Deviation); unit: mmol/mmol
Groups:
- Fasting: Fasting before surgery
- Water Group: Patients drank 800 ml of water 2 hrs before surgery
- Nutrition Group: Drank a carbohydrate drink 800 ml in the evening before surgery and 400 ml 2 hrs before surgery
Arm/Group | Fasting | Water Group | Nutrition Group
Number analyzed (Participants) | 20 | 19 | 18
mmol/mmol | 18.0 (2.0) | 17.3 (2.6) | 17.5 (2.7)

ADVERSE EVENTS:
Arm/Group | Fasting | Water | Carbohydrate Drink
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/18 | 0/19

LIMITATIONS AND CAVEATS:
A few glucose tolerance tests had to be discarded because of hemolysis in the samples taken for analysis of insulin.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No